CLINICAL TRIAL: NCT05588037
Title: Clinical Assessment of Combined Vitrectomy and Femtosecond Laser-assisted Cataract Surgery
Brief Title: Combined Vitrectomy and Femtosecond Laser-assisted Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHIRB2018019
Record Dates: First submitted 2020-12-08; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Macular Disease; Rhegmatogenous Retinal Detachment; Epiretinal Membrane; Cataract; Vitreous Hemorrhage; Vitreomacular Traction; Vitreous Cloudy
MeSH Terms: conditions — Macular Degeneration; Epiretinal Membrane; Cataract; Vitreous Hemorrhage | interventions — Air; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RRD group (Experimental): to evaluate the efficacy and complications of a new minimally invasive vitreoretinal surgery combined with FLACS in the treatment of rhegmatogenous retinal detachment complicated with cataract.
  Interventions: Procedure: FLACS +PPV+IOL + air
- ERM group (Experimental): to evaluate the efficacy and complications of a new minimally invasive vitreoretinal surgery combined with FLACS in the treatment of epiretinal membrane complicated with cataract.
  Interventions: Procedure: FLACS +PPV+IOL + epiretinal membrane peeling + Ozurdex
- MH group (Experimental): to evaluate the efficacy and complications of a new minimally invasive vitreoretinal surgery combined with FLACS in the treatment of macular hole complicated with cataract.
  Interventions: Procedure: FLACS + PPV+IOL + internal limiting membrane peeling + air
- Vitreous cloudy group (Experimental): to evaluate the efficacy and complications of a new minimally invasive vitreoretinal surgery combined with FLACS in the treatment of vitreous opacity complicated with cataract.
  Interventions: Procedure: FLACS + PPV+IOL

INTERVENTIONS:
Procedure: FLACS +PPV+IOL + air — The procedures are combined the FLACS +PPV+IOL + air.
  Arms: RRD group
Procedure: FLACS +PPV+IOL + epiretinal membrane peeling + Ozurdex — The procedures are combined the FLACS +PPV+IOL + epiretinal membrane peeling + Ozurdex.
  Arms: ERM group
Procedure: FLACS + PPV+IOL + internal limiting membrane peeling + air — The procedures are combined the FLACS + PPV+IOL + internal limiting membrane peeling + air.
  Arms: MH group
Procedure: FLACS + PPV+IOL — The procedures are combined the FLACS + PPV+IOL.
  Arms: Vitreous cloudy group

SUMMARY:
Based on the progress of cataract surgery, intraocular lens development, vitreoretinal surgery and anesthesia technology in recent years, the purpose of this study is to develop a new type of more accurate and minimally invasive combined surgery for cataract and fundus diseases, and to evaluate the advantages and value of the surgery as well as related complications, so as to minimize the surgical trauma and obtain faster visual function recovery and better patient comfort. To provide new solutions for the growing demand of eye health care.

DETAILED DESCRIPTION:
To evaluate the efficacy and complications of a new type of minimally invasive femtosecond laser assisted-cataract surgery (FLACS) combined with pars plana vitrectomy (PPV) with two-step anesthesia in the treatment of various common fundus diseases such as rhegmatogenous retinal detachment (RRD), epiretinal membrane (ERM), macular hole (MH), and vitreous opacity, complicated with cataract. It is mainly aimed at the following kinds of common fundus diseases with cataract performing PPV and cataract removal combined with monofocal or premium intraocular lens (IOL) implantation： RRD complicated with cataract: FLACS +PPV + IOL+air; ERM complicated with cataract: FLACS +PPV+IOL + epiretinal membrane peeling + Ozurdex; MH complicated with cataract: FLACS + PPV+ IOL + internal limiting membrane peeling + air; Vitreous opacity with cataract: FLACS + PPV+ IOL.

ELIGIBILITY:
Inclusion Criteria: clinical diagnosis of following disease

* RRD with cataract
* ERM with cataract
* MH with cataract
* Vitreous opacity with cataract

Exclusion Criteria: patients with history of following condition

* intraocular surgery
* ocular trauma
* endophthalmitis
* uveitis
* glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
visual acuity | Change from baseline best-corrected visual acuity at 6 months.
  final best-corrected visual acuity

SECONDARY OUTCOMES:
complications | through study completion, an average of 6 months.
  complications occurred during surgery or post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wensheng Li, Study Chair — Aier Ophthalmology School of Central South University; Shanghai Aier Eye Hospital
Locations (1):
- Jiasong Yang, Shanghai, China